CLINICAL TRIAL: NCT04592471
Title: Assessment of the Safety and Performance of Knee Ligament Supports in the Context of a Return to Sport After Sprain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Decathlon SE (Industry)
Collaborators: EFOR, France (Industry)
Responsible Party: Sponsor
Other Study IDs: kneeMID500-STRONG700
Record Dates: First submitted 2020-09-06; First posted 2020-10-19 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Knee Sprain (Mild); Knee Sprain (Moderate); Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Lymphoma, Follicular; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Orthosis Group 1: Use of kneeMID500 device
  Interventions: Device: kneeMID500-STRONG700
- Control Group 1: Control Group of the kneeMID500 Orthosis Group - No use of the device
- Orthosis Group 2: Use of kneeSTRONG700 device
  Interventions: Device: kneeMID500-STRONG700
- Control Group 2: Control Group of the kneeSTRONG700 Orthosis Group - No use of the device

INTERVENTIONS:
Device: kneeMID500-STRONG700 — At least 30 patients (15 patients in the orthosis group and 15 patients in the control group) per device type (2 device types: Knee MID 500 and Knee STRONG 700) totalling 60 patients will be included. Patients included in the orthosis group will use the device during sports sessions while patients included in the control group will not use a knee support device.
  Groups: Orthosis Group 1; Orthosis Group 2

SUMMARY:
Decathlon has developed kneeMID500-STRONG700 products which are two medical devices designed to be used for sport resumption after mild (kneeMID500) or moderate (KneeSTRONG100) knee sprain or after an Anterior Cruciate Ligament surgery.

The difference between these devices is based on the strength of compression and the knee maintain.

The objective of this multicentre study is to collect data on the related clinical complications and clinical outcomes of market-approved Decathlon kneeMID500-STRONG700 products to demonstrate safety and performance of these devices in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥18 years old
* Subject has a recent mild (grade I) OR moderate (grade II) knee sprain OR an ACL surgery
* The current condition of his/her knee allows the subject to resume usual physical activity
* Subject has been informed and is willing to sign an informed consent form
* Subject is willing to comply with protocol requirements and return to the study center for all clinical evaluations and required follow-up (18 weeks)
* Subject is affiliated to the French social security regime

Non-inclusion Criteria:

* Subject has conditions that may interfere with his/her ability to understand protocol requirements, participate in scheduled visits, or provide his/her informed consent
* Subject has worn a support (knee brace or articulated orthosis) since his/her recent injury
* Subject has resumed regular physical activity since his/her recent injury
* Subject has any medical condition that could impact the study at investigator's discretion
* Subject has a known hypersensitivity or allergy to the components of the device (polyamide, elastane, elastodiene)
* Adult subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with a recent mild (grade I) OR moderate (grade II) knee sprain OR an ACL surgery whose current condition of his/her knee allows the subject to resume usual physical activity.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Functional score | At baseline and 18 weeks of follow-up
  Comparison of the functional result (Lysholm Score: 0-100 points ; Tegner Activity Scale: 11-level gradient) between the baseline and last follow-up visit in each group (orthosis vs control), for each device model

SECONDARY OUTCOMES:
Confidence level | At baseline and 18 weeks of follow-up
  Gap in the confidence level (patient rated outcome with 6 questions, ranging from 0 to 100) related to physical activity, between the baseline and last follow-up visit in each group (orthosis vs control), for each device model
Knee instability | At 6 weeks, 12 weeks and 18 weeks of follow-up
  Comparison of knee instability, assessed through a numerical rating scale (NRS, ranging from 0 to 10), between the groups (orthosis vs control), for each device model
Knee pain | At 6 weeks, 12 weeks and 18 weeks of follow-up
  Comparison of knee pain, assessed through NRS (ranging from 0 to 10), between the groups (orthosis vs control), for each device model
Safety (adverse events) | 18 weeks of follow-up
  Comparison of adverse events rates between the groups (orthosis vs control), for each device model

CONTACTS AND LOCATIONS:
Overall Officials: Valérie WIECZOREK, Principal Investigator — Centre Hospitalier Universitaire de Lille
Locations (2):
- France (2):
  - Centre de rééducation et de balnéothérapie Kinés Faches, Faches-Thumesnil
  - Centre Hospitalier Universitaire de Lille, Lille

IPD SHARING:
Plan to Share IPD: No